CLINICAL TRIAL: NCT04559295
Title: Study of Bone of Marrow Concentrate (BMC) Injection in Discs, Facets, Sacroiliac Joints, and Epidural Space for Chronic Lower Back Pain With and Without Radiculopathy
Brief Title: Bone Marrow Concentrate (BMC) Injection in Intervertebral Discs
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stem Cures (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Regen_003-1018
Record Dates: First submitted 2020-08-31; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain; Disc Disease; Disc Degeneration; Arthropathy Vertebrae; Sacral Disorder; Radiculopathy; Spinal Stenosis
Keywords: Stem cells; Bone marrow concentrate; Disc; Minimally invasive; Injections; Facet joint; Sacroiliac joint; Epidural space
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration; Radiculopathy; Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: A prospective evaluation of a cohort of patients with a specific characteristic over time to see if they develop a particular endpoint or outcome based on a stated hypothesis.
Who Masked: Outcomes Assessor
Masking Description: Independent Observer was blinded as to wether a subject received treatment or was in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stem Cells (BMC) (Experimental): Subjects in the BMC arm received an injection of bone marrow concentrate
  Interventions: Biological: Bone Marrow Concentrate
- Control (No Intervention): Subjects in the control arm received no treatment for their condition

INTERVENTIONS:
Biological: Bone Marrow Concentrate — The intradiscal delivery of bone marrow concentrate (BMC) into discs, facet , epidural space, and sacroiliac joints
  Other Names: Stem Cells
  Arms: Stem Cells (BMC)

SUMMARY:
Intradiscal delivery of bone marrow concentrate (BMC) into discs, facet, epidural space, and sacroiliac joints

DETAILED DESCRIPTION:
To study if the outcomes for the injection of bone marrow concentrate (BMC) in patients with disc, facet, epidural space, and sacroiliac joint pain create a clinically meaningful improvement in pain and function. Further analysis will determine if there be any variance in patient reported outcome due to the individual's pre-procedure cell count and analysis.

Hypothesis 1: An injection of autologous BMC into discs, facets, sacroiliac joints, and epidural space will improve pain and function in patients with IDD

Hypothesis 2: There will be a direct relationship between an individual's BMC composition and the patient's reported outcomes

ELIGIBILITY:
Inclusion Criteria:

* A high index of suspicion for discogenic pain, i.e. painful degenerative discs with or without protrusions/herniations and facet/sacroiliac joint pain
* Patients with mild to severe spinal stenosis
* Patients with radiculopathy
* Patients with disc extrusions
* Patients with failed spinal fusion
* Patients with mild to severe facet arthropathy
* Patients with suspected sacroiliac joint disease
* Age 18 to 60 years
* Mild to severe loss of intervertebral disc height
* Pain is not responsive to conservative treatment measures (oral medication, epidural steroid injections, physical therapy)
* Pain persists for an extended period of time (i.e., at least 3 months)
* High intensity zone (HIZ) in annular fissure or adjacent to annular fissure detected on T2 or STIR MRI
* No evidence of contraindications to undergo procedure such as pregnancy, active infection, bleeding disorder, or metastatic cancer
* English speaking

Exclusion Criteria:

* Spinal Deformity (Scoliosis >20 degrees, Spondylolisthesis)
* Sequestered fragments, severe thecal sac compression
* Severe neurologic deficit
* Non-English speaking
* Bone marrow disorders
* Immunosuppressed Patients
* Patients with coagulopathy
* Localized infection in the area of skin penetration
* Spinal infection
* Serious medical co-morbidities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Two Years
  The Oswestry Disability Index (ODI) is a questionnaire used by clinicians and researchers to quantify disability for low back pain. Scale for the ODI is from 0 (best) - 100 (worst).

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | Two Years
  The NRS consists of a numeric version of the visual analog scale. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible. Scale for NRS is from 0 (best) - 10 (worst).
Visual Analog Scale (VAS) for back pain | Two Years
  When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. Scale for VAS for back pain is from 0 (best) - 10 (worst).
Visual Analog Scale (VAS) for leg pain | Two Years
  When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. Scale for VAS for leg pain is from 0 (best) - 10 (worst).
PROMIS Physical Health | Two Years
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. Scale for PROMIS Physical Health is from 16.2 (worst) - 67.7 (best)
PROMIS Mental Health | Two Years
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. Scale for PROMIS Mental Health is from 21.2 (worst) - 67.6 (best).
North American Spine Society (NASS) for patient satisfaction | Two Years
  The North American Spine Society (NASS) developed an outcome assessment instrument to measure diverse dimensions of the impact of lumbar spine problems. Scale range is from 1 to 4 (best to worst).
EURO Quality of Life (EuroQol) | Two Years
  EuroQol is an instrument which evaluates the generic quality of life developed in Europe and widely used. Scale is from 0.33 (worst - 0.88 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Atluri, MD, Principal Investigator — Stem Cures
Locations (1):
- Stem Cures, Cincinnati, Ohio, United States